CLINICAL TRIAL: NCT02916927
Title: Intravenous Sub-dissociative Dose Ketamine Injection Versus Infusion for Analgesia in the Emergency Department: A Prospective, Randomized, Double-blind Placebo Controlled Trial
Brief Title: Intravenous Sub-dissociative Dose Ketamine Injection Versus Infusion for Analgesia in the Emergency Department
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alameda Health System (Other)
Responsible Party: Principal Investigator, Eben Clattenburg, Investigator, Alameda Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00002
Record Dates: First submitted 2016-09-26; First posted 2016-09-28 (Estimated); Results first posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Pain
Keywords: ketamine; emergency department
MeSH Terms: conditions — Pain; Emergencies | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine IV infusion (Experimental): Ketamine 0.3 mg/kg in 100 mL normal saline minibag infused over 15 minutes. Placebo: 10 mL normal saline in syringe pushed over 1 minute. Masking: placebo normal saline minibags and placebo syringes will appear identical to the normal saline minibus and syringes with ketamine.
  Interventions: Drug: Ketamine IV Infusion
- Ketamine IV push (Active Comparator): Ketamine 0.3 mg/kg in a syringe pushed over 1 minutes. Placebo: 100 mL normal saline minibag infused over 15 minutes. Masking: placebo normal saline minibags and placebo syringes will appear identical to the normal saline minibus and syringes with ketamine.
  Interventions: Drug: Ketamine IV push

INTERVENTIONS:
Drug: Ketamine IV Infusion — Ketamine 0.3 mg/kg in 100mL normal saline minibag administered over 15 min and placebo 10 mL normal saline syringe administered over 1 minute.
  Other Names: Ketalar
  Arms: Ketamine IV infusion
Drug: Ketamine IV push — Ketamine 0.3 mg/kg in 10 mL normal saline syringe administered over 1 minute and placebo 100mL normal saline minibag administered over 15 min.
  Other Names: Ketalar
  Arms: Ketamine IV push

SUMMARY:
Objective: The purpose of this study is to determine if administering ketamine as an intravenous (IV) infusion over 15 minutes, as compared to an IV push, will decrease adverse drug reactions without attenuating its analgesic effects.

Study design: prospective, randomized, controlled, double-blind trial.

DETAILED DESCRIPTION:
Objective: The purpose of this randomized, controlled, double-blind trial is to evaluate if sub-dissociated dose ketamine given as an infusion versus an intravenous (IV) push over 1 minute has fewer and/or less severe adverse drug reactions and provides equivalent analgesia for patients with moderate to severe pain in the emergency department (ED).

Study design: Prospective, randomized, controlled, double-blind trial

Participants: Research assistants will recruit patients ≥18 years old with moderate to severe pain (NRS≥5) and an anticipated stay in the emergency department ≥1 hour. A sample size calculation was performed based on prior data which suggests that 60% of IV push arm and 20 % of infusion arm will have adverse drug reactions. investigators assume an alpha of 0.05 and a power of 0.8, which results in 56 patients needing to be enrolled.

Intervention: After a trained research assistant obtains written informed consent, pharmacists will randomize the participants to the IV push or IV infusion arm of the study. All patients will be placed on a cardiac monitor. All patients will receive and IV push over 1 minute and a 100 mL normal saline minibag over 15 minutes.

In the IV push arm, pharmacists will provide to the nurse ketamine 0.3 mg/kg in a 10 mL syringe and a 100 mL normal saline minibag. The nurse will start the minibag of normal saline and then administer the IV push of ketamine over 1 minute.

In the IV infusion arm, pharmacists will provide to the nurse ketamine 0.3 mg/kg in a 100 mL normal saline minibag and a 10 mL syringe of normal saline. The nurse will start the minibag of normal saline and then administer the IV push over 1 minute.

Data collection: The trained research assistant will collect data on the patients' pain scores, adverse drug reactions (presence, severity, and how bothersome they are), and vital signs.

Statistical analysis: Investigators will perform descriptive statistics, compare the proportion of patients with side effects, compare the severity of the side effects scores, and compare how bothersome the side effects.

ELIGIBILITY:
Inclusion Criteria:

* Pain NRS ≥5
* Anticipated stay in ED ≥1 hour

Exclusion Criteria:

* Pregnant or breast feeding
* Vital sign abnormalities (SBP <90, SBP > 180, HR < 50, HR > 150, RR <10, RR > 30, weight <45 kg, weight > 115 kg)
* Arrhythmias
* Altered mental status (active psychosis/delirium)
* Administration of opioid pain medication in previous 1 hour
* history of acute head or ocular trauma
* presence of known intracranial mass or vascular lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-09; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alameda Health System, Highland Hospital, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Clattenburg EJ, Hailozian C, Haro D, Yoo T, Flores S, Louie D, Herring AA. Slow Infusion of Low-dose Ketamine Reduces Bothersome Side Effects Compared to Intravenous Push: A Double-blind, Double-dummy, Randomized Controlled Trial. Acad Emerg Med. 2018 Sep;25(9):1048-1052. doi: 10.1111/acem.13428. Epub 2018 May 25. PMID 29645317

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 62 rather than 56 patients were enrolled because we were concerned about participants not completing the study.
Period: Overall Study
Arm/Group | Ketamine IV Infusion | Ketamine IV Push
Started | 31 | 31
Received Study Drug | 31 | 29
Completed | 30 | 28 (1 participant was in radiology for the 45 and 60 minute time points.)
Not Completed | 1 | 3
Not completed — Discharged prior to study drug receipt | 0 | 2
Not completed — At radiology for 45 & 60 min time points | 0 | 1
Not completed — Withdrawal before first time point | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine IV Infusion | Ketamine IV Push | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (12.0) | 46.6 (15.4) | 43.2 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 13 | 9 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Pain numeric rating scale at time 0 [Mean (Standard Deviation); unit: units on a scale] — Pain numeric rating scale (NRS) from 0 (no pain) to 10 (maximal pain).
  units on a scale | 8.6 (1.6) | 8.0 (1.4) | 8.3 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Side Effects
Description: The difference in percentage of participants endorsing side effects between each arm of the study over 60 minutes.
Time Frame: 0 - 60 minutes
Population: There are 30 rather than 31 participants in the ketamine IV infusion arm because one participant withdrew before the first time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine IV Infusion | Ketamine IV Push
Number analyzed (Participants) | 30 | 29
Participants | 21 | 25

2. Secondary Outcome: Side Effects
Description: The difference in percentage of participants endorsing side effects between each arm of the study at 5, 10, 15, 20, 30, 45, and 60 minutes.
Time Frame: 5, 10, 15, 20, 30, 45, 60 minutes
Population: 1 patient in the Ketamine IV push arm was in radiology for the 45 and 60 minute time points.
  There are 30 rather than 31 participants in the ketamine IV infusion arm because one participant withdrew before the first time point.
Measure: Number; unit: participants
Arm/Group | Ketamine IV Infusion | Ketamine IV Push
Number analyzed (Participants) | 30 | 29
participants
  5 minutes | 10 | 20
  10 minutes | 17 | 18
  15 minutes | 16 | 15
  20 minutes | 13 | 12
  30 minutes | 13 | 9
  45 minutes: number analyzed (Participants) | 30 | 28
  45 minutes | 9 | 5
  60 minutes: number analyzed (Participants) | 30 | 28
  60 minutes | 8 | 5

3. Secondary Outcome: Side Effect Severity
Description: The difference in severity of side effects (0 - 4) experienced by participants in each arm of the study at 5, 10, 15, 20, 30, 45, and 60 minutes. 0 indicates no side effects and 4 most severe side effects.
Time Frame: 5, 10, 15, 20, 30, 45, 60 minutes
Population: One patient in the Ketamine IV push arm was in radiology for the 45 and 60 minute time points.
  There are 30 rather than 31 participants in the ketamine IV infusion arm because one participant withdrew before the first time point.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ketamine IV Infusion | Ketamine IV Push
Number analyzed (Participants) | 30 | 29
units on a scale
  Fatigue at 5 minutes | 0.4 [0.03 to 0.8] | 0.6 [-0.05 to 1.1]
  Fatigue at 10 minutes | 0.9 [0.4 to 1.4] | 0.7 [0.3 to 1.2]
  Fatigue at 15 minutes | .6 [.2 to 1.0] | 0.7 [0.2 to 1.2]
  Fatigue at 20 minutes | 0.5 [-0.1 to 0.9] | 0.4 [0.1 to 0.8]
  Fatigue at 30 minutes | 0.2 [0.0 to 0.4] | 0.3 [-0.1 to 0.8]
  Fatigue at 45 minutes: number analyzed (Participants) | 30 | 28
  Fatigue at 45 minutes | 0.3 [-0.1 to 0.7] | 0.4 [-0.1 to 0.8]
  Fatigue at 60 minutes: number analyzed (Participants) | 30 | 28
  Fatigue at 60 minutes | 0.3 [-0.1 to 0.6] | 0.5 [0.0 to 0.9]
  Dizziness at 5 minutes | 0.8 [0.3 to 1.2] | 2.2 [1.6 to 2.9]
  Dizziness at 10 minutes | 1.1 [0.6 to 1.7] | 1.9 [1.3 to 2.5]
  Dizziness at 15 minutes | 1.1 [0.6 to 1.6] | 1.1 [0.6 to 1.7]
  Dizziness at 20 minutes | 1.0 [0.5 to 1.5] | 0.9 [0.5 to 1.3]
  Dizziness at 30 minutes | 0.4 [0.1 to 0.6] | 0.4 [0.1 to 0.8]
  Dizziness at 45 minutes: number analyzed (Participants) | 30 | 28
  Dizziness at 45 minutes | 0.2 [-01 to 0.5] | 0.3 [0.0 to 0.7]
  Dizziness at 60 minutes: number analyzed (Participants) | 30 | 28
  Dizziness at 60 minutes | 0.2 [-0.1 to 0.4] | 0.3 [0.0 to 0.7]
  Headache at 5 minutes | 0.2 [0.0 to 0.4] | 0.2 [-0.1 to 0.5]
  Headache at 10 minutes | 0.1 [0.0 to 0.2] | 0.3 [0 to 0.6]
  Headache at 15 minutes | 0.3 [0.0 to 0.6] | 0.3 [-0.1 to 0.6]
  Headache at 20 minutes | 0.2 [-0.1 to 0.5] | 0.2 [-0.1 to 0.5]
  Headache at 30 minutes | 0.3 [-0.1 to 0.7] | 0.2 [-0.1 to 0.5]
  Headache at 45 minutes: number analyzed (Participants) | 30 | 28
  Headache at 45 minutes | 0.2 [-0.1 to 0.5] | 0.3 [-0.1 to 0.6]
  Headache at 60 minutes: number analyzed (Participants) | 30 | 28
  Headache at 60 minutes | 0.2 [-0.1 to 0.5] | 0.3 [-0.1 to 0.6]
  Unreality at 5 minutes | 0.9 [0.4 to 1.4] | 2.6 [1.9 to 3.2]
  Unreality at 10 minutes | 1.5 [1.0 to 2.0] | 2.2 [1.6 to 2.8]
  Unreality at 15 minutes | 1.4 [0.9 to 1.9] | 1.3 [0.8 to 1.8]
  Unreality at 20 minutes | 1.1 [0.7 to 1.5] | 0.8 [0.4 to 1.1]
  Unreality at 30 minutes | 0.5 [0.2 to 0.8] | 0.2 [0.0 to 0.3]
  Unreality at 45 minutes: number analyzed (Participants) | 30 | 28
  Unreality at 45 minutes | 0.2 [-0.1 to 0.5] | 0.1 [0.0 to 0.2]
  Unreality at 60 minutes: number analyzed (Participants) | 30 | 28
  Unreality at 60 minutes | 0.1 [0.0 to 0.2] | 0 [0 to 0]
  Hearing at 5 minutes | 0.1 [-0.1 to 0.3] | 0.6 [0.1 to 1.1]
  Hearing at 10 minutes | 0.3 [0.0 to 0.7] | 0.2 [-0.1 to 0.5]
  Hearing at 15 minutes | 0.3 [0.0 to 0.7] | 0.2 [-0.1 to 0.5]
  Hearing at 20 minutes | 0.4 [0.0 to 0.8] | 0.1 [-0.1 to 0.3]
  Hearing at 30 minutes | 0.2 [-0.1 to 0.4] | 0.1 [-0.1 to 0.4]
  Hearing at 45 minutes: number analyzed (Participants) | 30 | 28
  Hearing at 45 minutes | 0 [0 to 0] | 0 [0 to 0]
  Hearing at 60 minutes: number analyzed (Participants) | 30 | 28
  Hearing at 60 minutes | 0 [0 to 0] | 0.04 [-0.02 to 0.05]
  Vision at 5 minutes | 0.03 [-0.03 to 0.1] | 0.7 [0.1 to 1.2]
  Vision at 10 minutes | 0.2 [0.0 to 0.4] | 0.4 [-0.1 to 0.8]
  Vision at 15 minutes | 0.2 [0.0 to 0.4] | 0.2 [-0.1 to 0.5]
  Vision at 20 minutes | 0.1 [-0.1 to 0.3] | 0.1 [-0.1 to 0.2]
  Vision at 30 minutes | 0.1 [-0.1 to 0.2] | 0.03 [-0.04 to 0.1]
  Vision at 45 minutes: number analyzed (Participants) | 30 | 28
  Vision at 45 minutes | 0 [0 to 0] | 0 [0 to 0]
  Vision at 60 minutes: number analyzed (Participants) | 30 | 28
  Vision at 60 minutes | 0 [0 to 0] | 0 [0 to 0]
  Mood at 5 minutes | 0.8 [0.3 to 1.3] | 1.7 [1.0 to 2.3]
  Mood at 10 minutes | 1.2 [0.7 to 1.7] | 2.3 [1.6 to 2.9]
  Mood at 15 minutes | 1.4 [0.9 to 1.8] | 2.0 [1.3 to 2.6]
  Mood at 20 minutes | 1.2 [0.8 to 1.7] | 1.2 [0.7 to 1.7]
  Mood at 30 minutes | 0.9 [0.5 to 1.3] | 0.6 [0.2 to 1.0]
  Mood at 45 minutes: number analyzed (Participants) | 30 | 28
  Mood at 45 minutes | 0.6 [0.2 to 1.0] | 0.3 [0.0 to 0.6]
  Mood at 60 minutes: number analyzed (Participants) | 30 | 28
  Mood at 60 minutes | 0.3 [0.1 to 0.6] | 0.1 [-0.1 to 0.3]
  Discomfort at 5 minutes | 0.1 [-0.1 to 0.3] | 0.4 [0.0 to 0.9]
  Discomfort at 10 minutes | 0.1 [0.0 to 0.2] | 0.4 [-0.1 to 0.9]
  Discomfort at 15 minutes | 0.1 [0.0 to 0.3] | 1.0 [0.8 to 1.9]
  Discomfort at 20 minutes | 0.2 [-0.1 to 0.4] | 0.4 [0.0 to 0.8]
  Discomfort at 30 minutes | 0.1 [0.0 to 0.3] | 0.3 [-0.1 to 0.6]
  Discomfort at 45 minutes: number analyzed (Participants) | 30 | 28
  Discomfort at 45 minutes | 0.2 [-0.1 to 0.4] | 0.2 [-0.1 to 0.5]
  Discomfort at 60 minutes: number analyzed (Participants) | 30 | 28
  Discomfort at 60 minutes | 0.2 [-0.1 to 0.5] | 0.3 [-0.1 to 0.7]
  Hallucinations at 5 minutes | 0.03 [0.0 to 0.1] | 0.9 [0.4 to 1.5]
  Hallucinations at 10 minutes | 0.1 [-0.1 to 0.2] | 0.7 [0.1 to 1.2]
  Hallucinations at 15 minutes | 0.03 [0.0 to 0.1] | 0.4 [0.0 to 0.7]
  Hallucinations at 20 minutes | 0.1 [-0.1 to 0.4] | 0.1 [0.0 to 0.2]
  Hallucinations at 30 minutes | 0.1 [-0.1 to 0.4] | 0 [0 to 0]
  Hallucinations at 45 minutes: number analyzed (Participants) | 30 | 28
  Hallucinations at 45 minutes | 0 [0 to 0] | 0 [0 to 0]
  Hallucinations at 60 minutes: number analyzed (Participants) | 30 | 28
  Hallucinations at 60 minutes | 0 [0 to 0] | 0 [0 to 0]

4. Secondary Outcome: How Bothersome Are the Side Effects?
Description: The difference in how bothersome (0, not bothersome, to 4, very bothersome, on the Side Effect Rating Scale for Dissociative Anesthetics "SERSDA") the side effects experienced by participants in each arm of the study are at 5, 10, 15, 20, 30, 45, and 60 minutes.
  "0" (no side effects), "1" (weak), "2" (moderate), "3" ("bothersome") to "4" (very bothersome)
Time Frame: 5, 10, 15, 20, 30, 45, 60 minutes
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Ketamine IV Infusion | Ketamine IV Push
Number analyzed (Participants) | 30 | 29
score on a scale
  Fatigue at 5 minutes | 0.1 [0.0 to 0.3] | 0.2 [-0.1 to 0.5]
  Fatigue at 10 minutes | 0.4 [0.1 to 0.8] | 0.3 [-0.1 to 0.7]
  Fatigue at 15 minutes | 0.3 [0.0 to 0.5] | 0.2 [-0.1 to 0.6]
  Fatigue at 20 minutes | 0.3 [0.0 to 0.6] | 0.2 [-0.1 to 0.5]
  Fatigue at 30 minutes | 0.1 [0.0 to 0.3] | 0.2 [-0.1 to 0.6]
  Fatigue at 45 minutes: number analyzed (Participants) | 30 | 28
  Fatigue at 45 minutes | 0.2 [-0.1 to 0.5] | 0.1 [-0.2 to 0.4]
  Fatigue at 60 minutes: number analyzed (Participants) | 30 | 28
  Fatigue at 60 minutes | 0.2 [-0.1 to 0.4] | 0.3 [-0.1 to 0.6]
  Dizziness at 5 minutes | 0.5 [0.1 to 0.9] | 1.4 [0.7 to 2.1]
  Dizziness at 10 minutes | 0.6 [0.2 to 1.1] | 0.9 [0.4 to 1.5]
  Dizziness at 15 minutes | 0.5 [0.1 to 0.9] | 0.7 [0.2 to 1.1]
  Dizziness at 20 minutes | 0.5 [0.0 to 0.9] | 0.6 [0.1 to 1.0]
  Dizziness at 30 minutes | 0.3 [0.0 to 0.6] | 0.2 [-0.1 to 0.5]
  Dizziness at 45 minutes: number analyzed (Participants) | 30 | 28
  Dizziness at 45 minutes | 0.2 [-0.1 to 0.4] | 0.2 [-0.1 to 0.5]
  Dizziness at 60 minutes: number analyzed (Participants) | 30 | 28
  Dizziness at 60 minutes | 0.2 [-0.1 to 0.4] | 0.2 [-0.1 to 0.5]
  Headache at 5 minutes | 0.2 [0.0 to 0.4] | 0.1 [-0.1 to 0.4]
  Headache at 10 minutes | 0.1 [0.0 to 0.2] | 0.2 [-0.1 to 0.6]
  Headache at 15 minutes | 0.2 [-0.1 to 0.5] | 0.3 [-0.1 to 0.7]
  Headache at 20 minutes | 0.1 [0.0 to 0.2] | 0.2 [-0.1 to 0.5]
  Headache at 30 minutes | 0.2 [-0.1 to 0.5] | 0.2 [-0.1 to 0.5]
  Headache at 45 minutes: number analyzed (Participants) | 30 | 28
  Headache at 45 minutes | 0.2 [-0.1 to 0.5] | 0.3 [-0.1 to 0.6]
  Headache at 60 minutes: number analyzed (Participants) | 30 | 28
  Headache at 60 minutes | 0.1 [0.0 to 0.3] | 0.2 [-0.1 to 0.5]
  Unreality at 5 minutes | 0.3 [0.0 to 0.6] | 1.6 [1.0 to 2.3]
  Unreality at 10 minutes | 0.6 [0.1 to 1.0] | 0.9 [0.4 to 1.5]
  Unreality at 15 minutes | 0.5 [0.1 to 1.0] | 0.4 [0.0 to 0.8]
  Unreality at 20 minutes | 0.5 [0.0 to 1.0] | 0.1 [0.0 to 0.2]
  Unreality at 30 minutes | 0.2 [-0.1 to 0.4] | 0.03 [0.0 to 0.1]
  Unreality at 45 minutes: number analyzed (Participants) | 30 | 28
  Unreality at 45 minutes | 0.1 [-0.1 to 0.4] | 0.03 [0.0 to 0.1]
  Unreality at 60 minutes: number analyzed (Participants) | 30 | 28
  Unreality at 60 minutes | 0.03 [0.0 to 0.1] | 0 [0 to 0]
  Hearing at 5 minutes | 0 [0 to 0] | 0.2 [-0.1 to 0.5]
  Hearing at 10 minutes | 0.2 [-0.1 to 0.4] | 0.1 [-0.1 to 0.4]
  Hearing at 15 minutes | 0.1 [-0.1 to 0.3] | 0.1 [0.0 to 0.2]
  Hearing at 20 minutes | 0.2 [-0.1 to 0.4] | 0.2 [-0.1 to 0.5]
  Hearing at 30 minutes | 0.1 [-0.1 to 0.2] | 0.1 [-0.1 to 0.4]
  Hearing at 45 minutes: number analyzed (Participants) | 30 | 28
  Hearing at 45 minutes | 0 [0 to 0] | 0 [0 to 0]
  Hearing at 60 minutes: number analyzed (Participants) | 30 | 28
  Hearing at 60 minutes | 0 [0 to 0] | 0.04 [0.0 to 0.1]
  Vision at 5 minutes | 0 [0 to 0] | 0.3 [-0.1 to 0.7]
  Vision at 10 minutes | 0.1 [-0.1 to 0.2] | 0.3 [-0.1 to 0.7]
  Vision at 15 minutes | 0.1 [-0.1 to 0.2] | 0.1 [-0.1 to 0.4]
  Vision at 20 minutes | 0.1 [-0.1 to 0.3] | 0.1 [-.01 to 0.4]
  Vision at 30 minutes | 0.1 [-0.1 to 0.4] | 0 [0 to 0]
  Vision at 45 minutes: number analyzed (Participants) | 30 | 28
  Vision at 45 minutes | 0 [0 to 0] | 0 [0 to 0]
  Vision at 60 minutes: number analyzed (Participants) | 30 | 28
  Vision at 60 minutes | 0 [0 to 0] | 0 [0 to 0]
  Mood at 5 minutes | 0.1 [-0.1 to 0.2] | 0.5 [0.0 to 0.9]
  Mood at 10 minutes | 0.2 [0.0 to 0.5] | 0.3 [0.0 to 0.6]
  Mood at 15 minutes | 0.2 [0.0 to 0.4] | 0.4 [0.0 to 0.8]
  Mood at 20 minutes | 0.2 [0.0 to 0.4] | 0.3 [-0.1 to 0.7]
  Mood at 30 minutes | 0.2 [0.0 to 0.5] | 0.03 [0.0 to 0.1]
  Mood at 45 minutes: number analyzed (Participants) | 30 | 28
  Mood at 45 minutes | 0.3 [-0.1 to 0.6] | 0 [0 to 0]
  Mood at 60 minutes: number analyzed (Participants) | 30 | 28
  Mood at 60 minutes | 0.1 [-0.1 to 0.4] | 0 [0 to 0]
  Discomfort at 5 minutes | 0.1 [-0.1 to 0.2] | 0.4 [0.0 to 0.9]
  Discomfort at 10 minutes | 0.1 [0.0 to 0.2] | 0.4 [-0.1 to 0.9]
  Discomfort at 15 minutes | 0.1 [0.0 to 0.2] | 0.4 [0.0 to 0.8]
  Discomfort at 20 minutes | 0.03 [0.0 to 0.1] | 0.4 [0.0 to 0.8]
  Discomfort at 30 minutes | 0.2 [-0.1 to 0.4] | 0.3 [-0.1 to 0.6]
  Discomfort at 45 minutes: number analyzed (Participants) | 30 | 28
  Discomfort at 45 minutes | 0.2 [-0.1 to 0.4] | 0.3 [-0.1 to 0.6]
  Discomfort at 60 minutes: number analyzed (Participants) | 30 | 28
  Discomfort at 60 minutes | 0.2 [-0.1 to 0.5] | 0.3 [-0.1 to 0.7]
  Hallucinations at 5 minutes | 0 [0 to 0] | 0.8 [0.2 to 1.3]
  Hallucinations at 10 minutes | 0.1 [-0.1 to 0.2] | 0.5 [0.0 to 0.9]
  Hallucinations at 15 minutes | 0 [0 to 0] | 0.3 [0.0 to 0.6]
  Hallucinations at 20 minutes | 0.1 [-0.1 to 0.4] | 0.1 [0.0 to 0.2]
  Hallucinations at 30 minutes | 0.1 [-0.1 to 0.4] | 0 [0 to 0]
  Hallucinations at 45 minutes: number analyzed (Participants) | 30 | 28
  Hallucinations at 45 minutes | 0 [0 to 0] | 0 [0 to 0]
  Hallucinations at 60 minutes: number analyzed (Participants) | 30 | 28
  Hallucinations at 60 minutes | 0 [0 to 0] | 0 [0 to 0]

5. Secondary Outcome: Reduction in Pain on Numeric Rating Scale.
Description: The difference in pain numeric rating score (NRS 0-10) experienced by participants in each arm of the study at 5, 10, 15, 20, 30, 45, and 60 minutes.
  Pain numeric rating scale from 0 (no pain) to 10 (maximal pain).
Time Frame: 5, 10 , 15, 20, 30, 45, 60 minutes
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Ketamine IV Infusion | Ketamine IV Push
Number analyzed (Participants) | 30 | 29
score on a scale
  5 minutes | 6.5 [5.4 to 7.7] | 2.9 [1.5 to 4.3]
  10 minutes | 5.4 [4.2 to 6.5] | 2.8 [1.5 to 4.1]
  15 minutes | 4.7 [3.6 to 5.7] | 3.4 [2.1 to 4.7]
  20 minutes | 4.3 [3.2 to 5.4] | 3.9 [2.7 to 5.1]
  30 minutes | 4.8 [3.8 to 5.9] | 4.2 [3.0 to 5.5]
  45 minutes: number analyzed (Participants) | 30 | 28
  45 minutes | 5.3 [4.3 to 6.3] | 4.6 [3.2 to 5.9]
  60 minutes: number analyzed (Participants) | 30 | 28
  60 minutes | 5.4 [4.4 to 6.5] | 4.5 [3.2 to 5.7]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the 60 minute study
Arm/Group | Ketamine IV Infusion | Ketamine IV Push
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/29
Other Adverse Events (participants affected / at risk) | 0/31 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-31): https://cdn.clinicaltrials.gov/large-docs/27/NCT02916927/Prot_SAP_000.pdf